CLINICAL TRIAL: NCT06954337
Title: MATCH-UP: MAking Telehealth-Delivery of Cancer Care at Home Effective and Safe-Upscaled: A Pragmatic Cluster Randomized Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-055
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: Telehealth; Cancer Care at Home; 25-055
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual practice pattern (UPP) (Active Comparator): Usual practice pattern (UPP) of patient's medical oncologist
  Interventions: Other: Usual practice pattern (UPP); Other: Experimental: Enhanced Telehealth (ET)
- Enhanced Telehealth (ET) (Experimental): Enhanced Telehealth (ET) practice pattern of patient's medical oncologist
  Interventions: Other: Usual practice pattern (UPP); Other: Experimental: Enhanced Telehealth (ET)

INTERVENTIONS:
Other: Usual practice pattern (UPP) — Patient follows usual practice pattern for routine care
Other: Experimental: Enhanced Telehealth (ET) — Patient follows enhanced telehealth practice pattern. As clinically appropriate, patients given option to shift routine care from face-to-face to at-home services available at institution: telehealth visits, home phlebotomy, and educational support for home administration of injection medications

SUMMARY:
Many people with cancer spend a lot of time and money traveling to and from the doctor's office for cancer care. MSK's goal is to make getting cancer care easier by cutting down the need to make in-person visits to MSK. MSK is trying to do this through a new option called enhanced telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast or prostate cancer at Memorial Sloan Kettering Cancer Center who have had at least 3 prior medical oncology visits.

Exclusion Criteria:

* Patient is enrolled on a therapeutic clinical trial.
* Patients whose primary language is not currently supported by Epic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of routine face to face medical oncology related visits out of total medical oncology related visits | 12 months
  all patients who meet eligibility criteria and have completed at least 2 medical oncology visits during the 12 month follow up period will be included for endpoint evaluability during analyses

CONTACTS AND LOCATIONS:
Overall Officials: Erin Bange, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm